CLINICAL TRIAL: NCT02736240
Title: Immunogenicity and Safety Study of the 13-valent Pneumococcal Polysaccharide Conjugate Vaccine Developed Cooperatively by YunNan Walvax Biotechnology Co., Lt and Yuxi Walvax Biotechnology Co., Lt Among 2-71 Months (the Youngest Could be 6 Weeks) Healthy Infants and Toddlers by Randomized Blind Method With Similar Control in Multi-centers.
Brief Title: Immunogenicity and Safety Study of the 13-valent Pneumococcal Polysaccharide Conjugate Vaccine in 2-71 Months Old Healthy Infants and Toddlers (the Youngest Could be 6 Weeks Old)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 022152015003
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Diseases Caused by Streptococcus Pneumoniae Serotypes
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Control Arm (Active Comparator): 7-valent pneumococcal conjugate vaccine
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine
- Test Arm (Experimental): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal polysaccharide conjugate vaccine

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugate vaccine
  Arms: Control Arm
Biological: 13-valent pneumococcal polysaccharide conjugate vaccine
  Arms: Test Arm

SUMMARY:
The purpose of this study is to investigate and valuate the immunogenicity and safety of the 13-valent pneumococcal polysaccharide conjugate vaccine in 2-71 months old healthy infants and toddlers (the youngest could be 6 weeks old)

ELIGIBILITY:
Inclusion Criteria:

* 2-71 months (the youngest could be 6 weeks old) infants or toddlers which are positively healthy based on the medical history, the physical examination and the judgment of the investigator;
* The statutory guardian (or the consignor) of the subject agree his/her child participate in the study, and is willing to sign the informed consent form;
* The subject and his/her statutory guardians (or the consignor) are able to comply with the requests of the clinical study protocol;
* Never be immunized with any pneumococcus vaccine, and didn't get immunization with any other preventive product in the past 10 days (didn't get immunized with attenuated live vaccine in the past 14 days);
* The auxillary temperature ≤37℃.

Exclusion Criteria:

* Has already been immunized with pneumococcus vaccine no matter it is experimental or marketed;
* With the history of invasive disease caused by streptococcus pneumonia by culture;
* With the history of serious allergy to any vaccine or drug, has got fever higher than 39℃ related to immunization with preventive biological product;
* Infant that the birth weight is lighter than 2.5 kg;
* With the history or the family history of seizure, epilepsy, cerebropathy and psychosis ;
* Infant with the abnormal labor (difficult labor, deliver with apparatus) or with the history of asphyxia or nervous damage;
* With the history of thrombocytopenia or other coagulation disorders by definite diagnosis;
* Infant or toddler with pathological jaundice by diagnosis;
* Be known with or suspected with immunological dysfunction, including immunosuppressive therapy (radiotherapy, chemotherapy, corticosteroid hormone, antimetabolites, cytotoxic drug), HIV infection etc. ;
* Be known with serious congenital malformation or serious chronic disease; suffer from congenital malformation or be diagnosed with serious chronic disease (eg. Down syndrome, diabetes mellitus, sickle cell anemia or nervous disease, Guillain-Barre syndrome);
* Be known with or suspected with diseases including: disease of respiratory system, acute infection or the active period of chronic disease, serious cardiovascular disease, hepatic-nephrotic disease, malignant tumor, skin disease;
* Has taken blood product or globulin (the hepatitis B immune globulin is allowed);
* Be participating in other clinical trials;
* Any other situation which is considered to influence the evaluation of the study by investigators .

Ages: 2 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2760 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-03 (Actual)

PRIMARY OUTCOMES:
positive rate after infant doses | 30 days after infant doses
  the rate of the immunoglobulin G ≥0.35μg/ml after infant doses
GMC after infant doses | 30 days after infant doses
  geometrical mean concentration of immunoglobulin G after infant doses
positive rate after booster dose | 30 days after booster dose
  the rate of the immunoglobulin G ≥0.35μg/ml after booster dose
GMC after booster dose | 30 days after booster dose
  geometrical mean concentration of immunoglobulin G after booster dose

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Principal Investigator — Beijing Chaoyang disease control and prevention center

REFERENCES:
- [Derived] Chen JJ, Yuan L, Huang Z, Shi NM, Zhao YL, Xia SL, Li GH, Li RC, Li YP, Yang SY, Xia JL. Safety and immunogenicity of a new 13-valent pneumococcal conjugate vaccine versus a licensed 7-valent pneumococcal conjugate vaccine: a study protocol of a randomised non-inferiority trial in China. BMJ Open. 2016 Oct 19;6(10):e012488. doi: 10.1136/bmjopen-2016-012488. PMID 27798013